CLINICAL TRIAL: NCT06761950
Title: Early Photobiomodulation Therapy on Pain and Range of Motion Following Flexor Tendon Repair
Brief Title: Photobiomodulation Therapy on Pain and Range of Motion Following Flexor Tendon Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rehab Hesham Mohamed El-Sheikh, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Reham-005391
Record Dates: First submitted 2024-12-31; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Photobiomodulation Therapy; Low Level Laser Therapy; Flexor Tendon Rupture; Flexor Tendon Repair
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Level Laser Therapy (Experimental): This group included 22 patients with zone II, and III flexor tendon injuries whom have pain and limited range of motion post flexor tendon repair surgery and received low-level laser therapy, 3 sessions per week, for a period of 4 weeks in addition to their physical therapy program and medical treatment
  Interventions: Device: Low Level laser therapy; Other: medical treatment; Other: physical therapy program
- placebo low level laser therapy (Active Comparator): This group included 22 patients with zone II, and III flexor tendon injuries whom have pain and limited range of motion after flexor tendon repair surgery and received placebo low-level laser therapy, 3 sessions per week for 4 weeks in addition to their physical therapy program and medical treatment.
  Interventions: Device: Placebo low level laser therapy; Other: medical treatment; Other: physical therapy program

INTERVENTIONS:
Device: Low Level laser therapy — The patient received low-level laser therapy three times per week for four weeks, with immobilization maintained. The Mustang 2000 Laser device was used with an infrared laser probe to accelerate tendon healing. The device's specifications include peak power output of 15W, power density of 15W/cm2, wave length of 890nm, pulse frequency of 100Hz, spherical size of 0.002cm2, pulse duration of 130 ns, exposure duration of 60 sec, and energy density of 5.85J/cm2.
  Arms: Low Level Laser Therapy
Device: Placebo low level laser therapy — Same as in the study group except turning on the device with covering probe by aluminum foil and ask patient to wear sun glasses to obtain the placebo effect 3 sessions per week for 4 weeks.
  Arms: placebo low level laser therapy
Other: medical treatment — the patients received their drugs from their treating physicians
Other: physical therapy program — patients received the traditional program after flexor tendon repair involving isometric exercise, stretching and mobilizations

SUMMARY:
The purpose of the study was to evaluate the therapeutic effect of low-level laser in improving pain and ROM following flexor tendon repair surgery.

DETAILED DESCRIPTION:
Flexor tendon injury is a common issue requiring early postoperative mobilization. Prolonged immobilization can lead to complications such as muscle atrophy, joint stiffness, osteoarthritis, infection, pain, joint cartilage ulceration, joint contracture, and tendon rupture. Low level laser therapy has been shown to accelerate inflammation, promote fibroblast proliferation, regulate procollagen messenger ribonucleic acid synthesis, accelerate bone repair and remodeling, encourage wound revascularization, and accelerate tissue repair. This study aims to evaluate the effectiveness of Low level laser therapy in pain management and improving range of motion after flexor tendon repair.

ELIGIBILITY:
Inclusion Criteria:

* Forty-four patients of both genders with age ranged between 20 to 50 years will participate in this study.
* All patients with zone II and III flexor tendon injuries, will be suffered from pain following flexor tendon repair surgery.
* All patients with zone II and III flexor tendon injuries, will be suffered from limitation of range of motion deficiency following flexor tendon repair surgery
* All patients enrolled to the study will have their informed consent.

Exclusion Criteria:

* A wound in the affected area
* Rheumatoid arthritis.
* Epilepsy or any psychological disorders
* Myelopathy or radiculopathy
* exposed hand tendons.
* Concomitant finger fractures, joint injuries, replantation or revascularizations, extensor tendon injury or crush injuries.
* Impairment of cognitive, perceptual or psychological function that would impede ability to follow verbal instruction.
* Multiple injuries to one flexor tendon, simultaneous injuries to bone and extensor tendons, skin loss, noncompliant patients or patients under 10 years, and gross contaminations of wounds.
* patients with tendon repair associated with a skin graft, nerve injury, arterial injury, systemic disease (e.g. diabetes mellitus), wound infection,

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-12-25 (Actual)

PRIMARY OUTCOMES:
Assessment of change of pain intensity | At baseline and after 4 weeks
  The Visual Analogue Scale is a 100mm line used for pain measurement, validated for various conditions like sleep, anxiety, breathlessness, and pruritus intensity. It accurately reflects pain changes, is reusable, and sensitive to acute pain changes.

SECONDARY OUTCOMES:
assessment of change of active range of motion of metacarpophalangeal joint | At baseline and after 4 weeks
  Goniometers, typically made of plastic or metal, measure the degree of motion in a single plane by aligning a stationary arm, a movable arm, and a fulcrum with the joint axis. it was used to measure the active range of motion of metacarpophalangeal joint when the patient is in a sitting position.
assessment of change of active range of motion of proximal interphalangeal joint | At baseline and after 4 weeks
  Goniometers, typically made of plastic or metal, measure the degree of motion in a single plane by aligning a stationary arm, a movable arm, and a fulcrum with the joint axis. it was used to measure the active range of motion of proximal interphalangeal joint when the patient is in a sitting position.
assessment of change of active range of motion of distal interphalangeal joint | At baseline and after 4 weeks
  Goniometers, typically made of plastic or metal, measure the degree of motion in a single plane by aligning a stationary arm, a movable arm, and a fulcrum with the joint axis. it was used to measure the active range of motion of distal interphalangeal joint when the patient is in a sitting position.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No